CLINICAL TRIAL: NCT03732729
Title: A Study for Evaluation of Massage Chair in Community-dwelling Older Adults: Randomized Study
Brief Title: Clinical Effect of Massage Chair on Older Adults
Acronym: SEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunju Lee (Other)
Collaborators: Bodyfriend (Unknown)
Responsible Party: Sponsor-Investigator, Eunju Lee, associate professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-1204
Record Dates: First submitted 2018-11-04; First posted 2018-11-07 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Older Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage chair (Experimental): lifestyle modification education(once)+ Using massage chair
  Interventions: Device: massage chair
- Control (No Intervention): lifestyle modification education(once)

INTERVENTIONS:
Device: massage chair — Patient should use massage chair, twice per day, for 30minutes
  Arms: Massage chair

SUMMARY:
The use of massage chairs is becoming more popular in many countries. According to the previous reports, some manual massages have positive effects on the mood, pain, fatigue, and sleep quality. However, the clinical benefits of the massage chair have not been fully understood. In this trial, it is aimed to evaluate the clinical effectiveness of the 6-month regular use of massage chair twice a day. It is hypothesized that long-term regular use of massage chair has positive effects on the hormonal level related to the stress, inflammation, and aging, as well as physical, psychologic, and muscle quality.

DETAILED DESCRIPTION:
A total of enrolled 80 patients after randomization(1:1) in intervention(Massage chair)group and Control groups, will be provided

* Massage chair group

  * lifestyle modification education + using massage chair twice per day during 24weeks
* control group: only lifestyle modification education

  1. Screening visit

     * collection demographic data, BMD, vital sign, Medication history
  2. Visit 1 (0-week)

     1. Vital sign
     2. Charlson comorbidity index
     3. Laboratory test

        * WBC diff count, Hb, creatinine, ALT, albumin, hsCRP, ESR cortisol, serotonin, DHEA-s, IGF-1, NK cell, Telomere length
     4. Questionnaire: K-MMSE, SGDS-K, BEPSI-K, EQ-5D-5L
     5. Physical& muscular assessment

        * SPPB, Grip strength, Muscle tone, Bioimpedance analysis
  3. Visit 2-6 (4,8,12,16 weeks) via Phone contact: assess compliance and adverse events
  4. visit 7 (24weeks)

     1. Vital sign
     2. Laboratory test

        * WBC diff count, Hb, creatinine, ALT, albumin, hsCRP, ESR cortisol, serotonin, DHEA-s, IGF-1, NK cell, Telomere length
     3. Questionnaire: K-MMSE, SGDS-K, BEPSI-K, EQ-5D-5L
     4. Physical& muscular assessment

        * SPPB, Grip strength, Muscle tone, Bioimpedance analysis
     5. Compliance
     6. Adverse events

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling healthy adults between 50-75 years old

Exclusion Criteria:

1. Unable to sign his/her own informed consent
2. Any disability or damages in 4 extremity.
3. Who have exercised regularly more than twice a week during the last 24 weeks
4. Who have received regular massage during the last 24 weeks
5. Confirmed osteoporosis of T score <-2.5 from BMD or history of compression fracture
6. Cortisol-metabolism disorders or other diseases that can affect steroid secretion
7. Who have taken any medication related with steroid secretion or metabolism within 2 weeks
8. Expected life expectancy less than 12 months (Symptomatic heart failure, end-stage renal failure)
9. Spouse is already enrolled in this research

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Serum cortisol level | Change from baseline serum cortisol level at 24weeks
  Investigate serum cortisol level of baseline & 24weeks between 2 groups.

SECONDARY OUTCOMES:
Cortisol/DHEA-s ratio | Change from Baseline cortisol/DHEA-s ratio level at 24weeks
  Investigate serum Cortisol/DHEA-s ratio level of baseline & 24weeks between 2 groups.
Serum Serotonin level | Change from Baseline serum serotonin level at 24weeks
  Investigate serum serotonin level of baseline & 24weeks between 2 groups.
Serum IGF-1 level | Change from Baseline Serum IGF-1 level level at 24weeks
  Investigate serum IGF-1 level of baseline & 24weeks between 2 groups.
ESR | Change from Baseline ESR level at 24weeks
  Investigate serum ESR level of baseline & 24weeks between 2 groups.
hsCRP | Change from Baseline hs CRP level at 24weeks
  Investigate serum hsCRP level of baseline & 24weeks between 2 groups.
NK cell activity | Change from Baseline NK cell activity level at 24weeks
  Investigate serum NK cell activity of baseline & 24weeks between 2 groups.
Telomere length | Change from Baseline Telomere length level at 24weeks
  Investigate Telomere length of baseline & 24weeks between 2 groups
Korean version Short form Geriatric Depression Scale(SGDS-K) score | SGDS-K summed total score is changed lower at 24weeks from baseline
  15 item measure to assess the depression
Korean version -Brief Encounter Psychosocial Instrument(BEPSI-K) score | BEPSI-K summed total score is changed lower at 24weeks from baseline
  5 item measure to assess the Stress
The 5-level EQ-5D version(EQ-5D-5L) score | EQ-5D-5L summed total score is changed higher at 24weeks from baseline
  6 item measure to assess the quality of life
Muscle tone score | Individual site Muscle tone score is changed higher at 24weeks from baseline
  6 item measure to assess Muscle tone of both trapezoid& forearm & thigh

CONTACTS AND LOCATIONS:
Overall Officials: Eunju Lee, Principal Investigator — Asan Medical Center
Locations (1):
- AsanMC, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No